CLINICAL TRIAL: NCT01912274
Title: A Phase II Open-Label, Single-arm, Two-Stage, Multicenter Trial of Pracinostat in Combination With Azacitidine in Elderly (Age 65 Years or Older) Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Safety and Efficacy Study of Pracinostat With Azacitadine in Elderly Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEI-004
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; open label; nonrandomized; single arm; elderly patients; HMA; newly diagnosed
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SB939 compound; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pracinostat with azacitadine (Experimental): 60 mg of pracinostat by mouth 3 times a week for 3 weeks followed by 1 week of rest repeated every 28 days 75 mg/m2 azacitadine for the first 7 days of each 28 day cycle, via subcutaneous (SC) injection or intravenous (IV) infusion if SC injections are intolerable
  Interventions: Drug: Pracinostat; Drug: Azacitidine

INTERVENTIONS:
Drug: Pracinostat — Elderly newly diagnosed patients will all receive pracinostat
  Other Names: SB939
Drug: Azacitidine — Elderly newly diagnosed patients will all receive azacitadine
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of pracinostat when combined with azacitadine for patients who are 65 years of age or older and have Acute Myelogenous Leukemia (AML)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥65 years.
* Voluntary written informed consent before performance of any study related procedure not part of normal medical care.
* Newly diagnosed de novo, secondary, or treatment-related AML with intermediate or unfavorable-risk cytogenetics based on the Southwest Oncology Group (SWOG) classifications (Slovak et al, 2000).
* One prior cycle of therapy with an approved hypomethylating agent (HMA) such as azacitidine or decitabine is allowed for either an antecedent hematologic disorder (AHD) or AML. Patients are also eligible if they have received lenolidamide, immunosuppressive therapy or low dose chemotherapy for their AHD. Prior hydroxyurea is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* ≥20% blasts in bone marrow.
* Peripheral WBC <30,000/uL.
* Adequate organ function as evidenced by:
* Total bilirubin 2x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)2.5x ULN
* Serum creatinine 2x ULN
* QT interval corrected according to Fridericia's formula (QTcF) ≤450 milliseconds (ms) for male subjects or ≤470 ms for female subjects on ECG at Screening.
* Male subjects who are surgically sterile or willing to use adequate contraceptive measures or abstain from heterosexual intercourse during the entire study treatment period.
* Female subjects who are not of childbearing potential.
* Willingness and ability to understand the nature of this study and to comply with the study and follow up procedures

Exclusion Criteria:

* Acute promyelocytic leukemia (French-American-British [FAB] M3 classification).
* Known AML-associated t(15;17), t(8;21), t(16;16), del(16q), or inv(16) karyotype abnormalities.
* Presence of a malignant disease within the last 12 months, with the exception of adequately treated in-situ carcinomas, basal or squamous cell carcinoma, or non-melanomatous skin cancer. Other malignancies will be considered on a case-by-case basis.
* Life-threatening illnesses other than AML, uncontrolled medical conditions or organ system dysfunction that, in the Investigator's opinion, could compromise the subject's safety, or put the study outcomes at risk.
* Uncontrolled or symptomatic arrhythmias, unstable angina, or any Class 3 or 4 cardiac diseases as defined by the New York Heart Association (NYHA) Functional Classification.
* Clinical evidence of central nervous system (CNS) involvement.
* Are candidates for intensive chemotherapy (induction chemotherapy, bone marrow, or stem cell transplant) within the next 4 months.
* Received more than one prior cycle of HMA, previous bone marrow transplant or other intensive chemotherapy regimens for either an AHD or AML.
* Received prior radiation therapy for extramedullary disease within 2 weeks of study enrollment.
* Received prior histone deacetylase (HDAC) inhibitor or deacetylase (DAC) inhibitor is not permitted such as Istodax (romidepsin/depsipetide) or valproic acid.
* Received hematopoietic growth factors: erythropoietin, granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), or thrombopoietin receptor agonists within 7 days (14 days for Aranesp) prior to study enrollment.
* Have been treated with any chemotherapeutic agent within 2 weeks or 5 half-lives of the first dose of study drug, whichever is longer.
* Are being treated with systemic corticosteroids. Inhaled and topical steroids as well as intermittent dexamethasone for nausea or vomiting are permitted.
* Known history of human immunodeficiency virus (HIV) or active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).
* Uncontrolled active systemic infections.
* Gastrointestinal (GI) tract disease, causing the inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, or uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis).
* Any disease(s), psychiatric condition, metabolic dysfunction, or findings from a physical examination or clinical laboratory test result that would cause reasonable suspicion of a disease or condition, that contraindicates the use of study drugs, that may increase the risk associated with study participation, that may affect the interpretation of the results, or that would make the subject inappropriate for this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12-24 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (17):
- United States (17):
  - City of Hope Comprehensive Cancer Ctr, Duarte, California
  - USC Norrris Cancer Center, Los Angeles, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Stanford University School of Medicine, Stanford, California
  - Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Inidana Univ Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Mercy Medical Research Center, Springfield, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Hospital, Camden, New Jersey
  - Oregon Health and Science University, Portland, Oregon
  - Medical College of South Carolina-Hollings Cancer Ctr, Charleston, South Carolina
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Medical College of Wisconsin-Froedtert Cancer Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Garcia-Manero G, Abaza Y, Takahashi K, Medeiros BC, Arellano M, Khaled SK, Patnaik M, Odenike O, Sayar H, Tummala M, Patel P, Maness-Harris L, Stuart R, Traer E, Karamlou K, Yacoub A, Ghalie R, Giorgino R, Atallah E. Pracinostat plus azacitidine in older patients with newly diagnosed acute myeloid leukemia: results of a phase 2 study. Blood Adv. 2019 Feb 26;3(4):508-518. doi: 10.1182/bloodadvances.2018027409. PMID 30760466
- See also: Sponsor website — http://www.meipharma.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pracinostat With Azacitadine
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 50
Age, Continuous [Median (Full Range); unit: years] | 75 [66 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Best Response Rate
Description: Proportion of patients assessed as having achieved a disease response of either CR or CRi or MLFS according to the IWG criteria. CR (ie, complete remission defined as <5% blasts in the bone marrow, no blasts with Auer rods, no extramedullary disease, ANC ≥1000/μL, and platelets ≥100,000/μL must be independent of transfusions for at least 1 week before each assessment).
  CRi (ie, morphologic complete remission with incomplete blood count recovery, defined as morphologic CR with residual neutropenia (<1,000/μL) or residual thrombocytopenia (<100,000/μL), no extramedullary disease, does not require transfusion independence) MLFS (ie, morphologic leukemia free state, defined as <5% blasts in an aspirate sample with marrow spicules, no extramedullary disease, does not require transfusion independence)
Time Frame: through study completion up to a maximum of three years
Population: ITT set
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 50
Participants | 26

2. Secondary Outcome: Overall Response Rate
Description: proportion of patients with CR plus CRi plus MLFS plus PR plus PRi
Time Frame: through study completion up to a maximum of three years
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 50
Participants | 32

3. Secondary Outcome: Complete Cytogenetic Response Plus Molecular Complete Remission
Description: proportion of patients assessed as having complete cytogenetic response (CRc) + molecular complete remission (CRm) to pracinostat plus azacitidine
Time Frame: through study completion up to a maximum of three years
Population: 17 patients had molecular abnormalities identified at baseline and were evaluable for assessing CRm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 17
Participants | 1

4. Secondary Outcome: Progression Free Survival
Description: time from the first day of study administration to PD, relapse from CR/CRi/MLFS, lack of efficacy or death.
Time Frame: through study completion up to a maximum of three years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 50
months | 12.56 [10.03 to 17.70]

5. Secondary Outcome: Overall Survival
Description: time from the first day of study drug administration to death
Time Frame: through study completion up to a maximum of three years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 50
months | 19.08 [10.00 to 26.52]

6. Secondary Outcome: Duration of Best Response
Description: The duration of the best response to treatment with pracinostat plus azacitidine was determined by the Investigator for patients who achieved a CR, CRi, or MLFS. The duration was defined as the time from the initial determination of response to the time of relapse, PD, or death, whichever occurred first plus 1 day.
Time Frame: through study completion up to a maximum of 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 26
months | 11.54 [8.30 to 17.18]

7. Secondary Outcome: Duration of Response
Description: The duration of the response to treatment with pracinostat plus azacitidine was determined by the Investigator for patients who achieved a CR, CRi, PR, PRi, or MLFS. The duration was defined as the time from the initial determination of response to the time of relapse, PD, or death, whichever occurred first plus 1 day.
Time Frame: through study completion up to a maximum of three years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pracinostat With Azacitadine
Number analyzed (Participants) | 32
months | 11.54 [8.30 to 17.18]

ADVERSE EVENTS:
Time Frame: through study completion up to a maximum of three years
Arm/Group | Pracinostat With Azacitadine
Serious Adverse Events (participants affected / at risk) | 50/50
Other Adverse Events (participants affected / at risk) | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pracinostat With Azacitadine (N=50)
pneumonia (Infections and infestations) | 3
sepsis (Infections and infestations) | 3
diverticulitis (Infections and infestations) | 2
enterococcal bacteraemia (Infections and infestations) | 2
oral infection (Infections and infestations) | 2
pseudomonal bacteraemia (Infections and infestations) | 2
septic shock (Infections and infestations) | 2
urinarytract infection (Infections and infestations) | 2
anal abscess (Infections and infestations) | 1
device relatedinfection (Infections and infestations) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Neutropenic sepsis (General disorders) | 1
Parainfluenzae virus infection (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia fungal (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
febrile neutropenia (Cardiac disorders) | 16
thrombocytopenia (Blood and lymphatic system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 1
headache (Nervous system disorders) | 1
cellulitis (Infections and infestations) | 4
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Cardiac tamponade (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Fatigue (General disorders) | 2
Pyrexia (Skin and subcutaneous tissue disorders) | 1
Systemic inflammatory response syndrome (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Laryngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1
Renal failure acute (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pracinostat With Azacitadine (N=50)
Nausea (Gastrointestinal disorders) | 24
Vomiting (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 20
Asthenia (General disorders) | 7
Chills (General disorders) | 5
Pyrexia (Hepatobiliary disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Neutropenia (Blood and lymphatic system disorders) | 15
Anaemia (Blood and lymphatic system disorders) | 11
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 4
Weight decreased (Investigations) | 6
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 3
Neuropathy peripheral (Nervous system disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 11
Pneumonia (Infections and infestations) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Contusion (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No